CLINICAL TRIAL: NCT06194201
Title: A Multi-centre, Randomized, Double-blind, Active Controlled, Parallel Groups, Phase II Study to Evaluate the Efficacy and Safety of Intravenous HRS9432 in the Treatment of Subjects With Candidemia and/or Invasive Candidiasis
Brief Title: A Trial of Intravenous HRS9432 in the Treatment of Subjects With Candidemia and/or Invasive Candidiasis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS9432-201
Record Dates: First submitted 2023-12-21; First posted 2024-01-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-12

CONDITIONS: Patients With Candidemia and/or Invasive Candidiasis
MeSH Terms: interventions — Caspofungin; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS9432 (Experimental)
  Interventions: Drug: HRS9432
- Caspofungin Acetate for Injection (Active Comparator)
  Interventions: Drug: Caspofungin Acetate for Injection

INTERVENTIONS:
Drug: HRS9432 — Dosing frequency: intravenously once week
  Arms: HRS9432
Drug: Caspofungin Acetate for Injection — Dosing frequency: D1 70mg，followed by 50mg intravenously once daily
  Arms: Caspofungin Acetate for Injection

SUMMARY:
The Purpose of this study is to evaluate the efficacy and safety of intravenous HRS9432 in patients with candidemia and/or invasive candidiasis

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥18 years；
2. Established or clinical diagnosis of candidemia and/or IC ；
3. Present of 1 or more systemic signs attribute to candidemia and/or IC 4 days prior to randomization;
4. Women of childbearing potential or male subjects whose partner is a fertile female agree to use highly effective form of contraception from the time of signed ICF till 6 months after end of treatment；
5. Able and willing to provide a written informed consent

Exclusion Criteria:

1. Any of the following forms of IC: including osteomyelitis, endocarditis or myocarditis, meningitis, endophthalmitis, or any central nervous system infection, urinary tract infection or chronic disseminated candidiasis；
2. Severe hepatic impairment in subjects with a history of chronic cirrhosis；
3. History of severe ataxia, tremor, or neuropathy or a diagnosis of multiple sclerosis or a movement;
4. Laboratory abnormalities in baseline specimens obtained at screening;
5. ECG with clinical significance and may cause obvious safety risk to the subjects at screening;
6. Received systemic treatment with an antifungal agent at approved doses for treatment of candidemia or IC for >48 hours;
7. Vascular catheter or device that cannot be removed, or abscess that cannot be drained, and may be the source of candidemia or IC;
8. A history of drug use, alcohol, or drug abuse within 1 year prior to randomization;
9. Participated in, any other clinical study involving the administration of active investigational or experimental medication prior to the randomization, or 5 half-lives, whichever is longer, prior to Screening;
10. Females who are in gestation or lactating period or planned pregnancy during the study
11. Known history of hypersensitivity or allergic reaction to HRS9432, caspofungin etc echinocandins drugs;
12. In the judgment of the Investigator, other reasons unsuitable for study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate overall success (mycological eradication and resolution of systemic signs attributable to candidemia and/or invasive candidiasis [IC]) of HRS9432 IV in subjects with candidemia and/or IC in the Microbiological Intent-to-treat (mITT) population | Day 14

SECONDARY OUTCOMES:
Evaluate overall success (mycological eradication and resolution of systemic signs attributable to candidemia and/or IC) of HRS9432 IV in the mITT population | Day 5, Day 28, End of treatment(≤2 days of last dose) and End of Study (Day 56±3 days)]
Evaluate clinical cure as assessed by the Investigator for HRS9432 IV in the mITT population | Day 5, Day 14, Day 28, End of Treatment (≤2 days of last dose) and End of Study (Day 56±3 days)
Evaluate mycological success(eradication) of HRS9432 IV in the mITT population | Day 5, Day 14, Day 28, End of Treatment (≤2 days of last dose) and End of Study (Day 56±3 days)
Evaluate All cause Mortality in the mITT population | Day 28 and End of Study (Day 56±3 days)
The time when two consecutive negative candida cultures occurred for the first time with an interval of ≥12h in the mITT population | Day1 through End of Study (Day 56±3 days)
Percentage of Participants with mycological recurrence in the mITT population | End of Treatment (≤2 days of last dose) andEnd of Study (Day 56±3 days)
Time of the first mycological recurrence in the mITT population | Day1 through End of Study (Day 56±3 days
Number of Participants With Adverse Events and severity | Day1 through End of Study (Day 56±3 days)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital Of University Of South China, Hengyang, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided